CLINICAL TRIAL: NCT06102655
Title: Effect and Mechanism of Jiajian Guishen Formulation on Premature Ovarian Insufficiency
Brief Title: Effect and Mechanism of Jiajian Guishen Formulation on Premature Ovarian Insufficiency Based on Metabolomics
Acronym: JJGS and POI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shi Yun (Other)
Responsible Party: Sponsor-Investigator, Shi Yun, Sponsor-Investigator, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023DZMEC-290; 2023DZMEC-290-02 (Other: Ethics Committee of Dongzhimen Hospital Affiliated to Beijing University of Chinese Medicine)
Record Dates: First submitted 2023-10-18; First posted 2023-10-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-09

CONDITIONS: Premature Ovarian Insufficiency; Metabolomics; Traditional Chinese Medicine; Mechanism; Clinical Syndrome
Keywords: Premature Ovarian Insufficiency; Metabolomics; Traditional Chinese Medicine; Mechanism; Clinical Syndrome
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group（Jiajian Guishen Formulation） (Experimental): Jiajian Guishen Formulation is a traditional Chinese medicine, it will be used in POI patients for three menstrual cycles; their blood samples are collected before and after treatment.
  Interventions: Drug: Jiajian Guishen Formulation
- no-treatment control group (No Intervention): healthy people

INTERVENTIONS:
Drug: Jiajian Guishen Formulation — Jiajian Guishen Formulation is a formulation of Traditional Chinese Medicine.POI patients will be treat with Jiajian Guishen Formulation for three menstrual cycles; their blood samples are collected before and after treatment.No drug will be used in control group, and their blood samples are collected when join the experiment.
  Arms: treatment group（Jiajian Guishen Formulation）

SUMMARY:
1. Identify differential metabolites in POI patients.
2. Analysis of differential metabolites and their involved mechanism pathways.

ELIGIBILITY:
Inclusion Criteria:

POI Inclusion Criteria:

1. Patients diagnosed by Western medicine with premature ovarian insufficiency;
2. Patients with Chinese medicine differentiation of kidney deficiency and liver depression;
3. 18 ≤ patients' age ≤ 39 years;
4. Patients who do not use other drugs during treatment;
5. Patients who voluntarily participate in this study, sign an informed consent form, and agree to take the corresponding treatment plan.

The above five items must be met to be included in the POI patient group in this study.

Healthy subjects inclusion criteria:

1. 18 ≤ Age≤ 39 years old;
2. menstrual regularity;
3. There is no abnormality in sex hormone and AMH examination;
4. Voluntarily participate in this research and sign the informed consent form;
5. Those who match the general information such as age, height, and weight of the patients included in POI.

Exclusion Criteria:

POI exclusion criteria:

1. Patients with congenital gonadal dysplasia or a family history similar to "early menopause";
2. POI patients with acquired organic lesions or ovarian surgery;
3. Patients who have taken Western medicine artificial cycle therapy or other endocrine therapy in the past three months;
4. Patients with serious primary diseases and mental disorders such as cardiovascular and cerebrovascular, liver, kidney and hematopoietic system;
5. Patients who are breastfeeding or pregnant;
6. Patients who are allergic to the drugs used in this study or have a history of previous allergy to traditional Chinese medicines.

Those who met any of the above 5 criteria were excluded from this study. Healthy subjects were excluded as (1), (3), (4), (5).

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — biological
Enrollment: 46 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
follicle stimulating hormone,FSH | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.

SECONDARY OUTCOMES:
anti mullerian hormone, AMH | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
Evaluation of the efficacy of Traditional Chinese Medicine symptoms | before and1 month after the treatment
  A sacle score to evalyate the symptoms, results of scores ranges from 0 to 108, higher scores mean more severe condition of POI.The main symptoms include menstrual cycle, menstrual flow reduction. Scoring criteria: ① normal menstrual cycle 0 points, 1-2 weeks ahead or behind the wrong 4 points, 2-3 weeks 8 points, more than 3 weeks 12 points; ② menstrual flow than the previous menstrual flow no change 0 points, menstrual flow reduction ≤ ⅓ 4 points, ⅓ < menstrual flow reduction ≤ ½ 8 points, menstrual flow reduction > ½ 12 points. Secondary symptoms included lumbar and knee pain, dizziness and tinnitus, loss of libido, increased urination, hot flashes and night sweats, and lower back and lower limb pain et. According to the degree of aggravation of symptoms, the total score was assigned as 0,2,4,8.
Improved Kupperman Scale Scoring | before and 1 month after the treatment
  A sacle score to evalyate the symptoms, results of scores ranges from 0 to 39, higher scores mean more severe condition of POI.Referring to the domestic modified Kupperman Symptom Scoring Criteria in Chinese Obstetrics and Gynecology, edited by Cao Zeyi, to observe and rate perimenopausal symptoms before and after treatment and to quantify the degree of decline in ovarian function.Entries include hot flashes and sweating, sensory abnormalities, insomnia, anxiety and depression, dizziness, fatigue, muscle and joint pain, headache, palpitations, ankylosis of the skin, sexual discomfort, and urinary irritation, with different coefficients for each entry, and according to the aggravating degree of the symptom, they are divided into 0, 1, 2, and 3 points, and the coefficients corresponding to the scoring of the degree of each item are multiplied by a fixed score of the symptom to add up to the total score.
estradiol, E2 | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
luteinizing hormone, LH | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
testosterone, T | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
malondialdehyde | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
superoxide dismutase | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
reduced glutathione, GSH | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
ceruloplasmin | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
copper | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
metabolite level | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment.
Differential metabolites and their related indexes of mechanism pathways | Differential metabolites will be tested on the 2~4th day of menstruation (amenorrhea patients before and after taking medication), related indexes of mechanism pathways will be tested after the analyses of differential metabolities
  The results of differential metabolites and their related indexes of mechanism pathways cann't be predicted until the metabolomics test finish, because the test include hundreds of metabolites. Metabolomics results will be tested by using liquid chromatography coupled with mass spectrometry (LC-MS) to identify potential markers.All multivariate analyses and modeling on the normalized data were carried out using software SIMCA-P. Supervised analysis (orthogonal partial least squares discriminate analysis, OPLS-DA) was applied to distinguish metabolic difference between normal group and POI group. SPSS 22.0 (SPSS Inc) software was used for receiver operating characteristic (ROC) curve analyses and binary logistic regression analyses. Then their related indexes of mechanism pathways will be tested in blood samples.
Number of participants with abnormal laboratory test of blood routine examination results | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment. white blood cell count (WBC), red blood cell (RBC) and platelet count/blood platelet count (PLT) are included.
Number of participants with abnormal Liver and kidney function (by laboratory test results) | On the 2~4th day of menstruation (amenorrhea patients before and after taking medication)
  Blood samples are collected before and after treatment. creatinine(CREA), uric acid (UA), alanine amiotransferase(AST), aspartate aminotransferase (AST) and γ-glutamyl transpeptadase (GGT) are included.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Shi, Study Director — Dongzhimen Hospital of Beijing University of Chinese Medicine; Ke Xu, Master, Principal Investigator — Dongzhimen Hospital of Beijing University of Chinese Medicine; Jing yi Shao, Master, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine; Xi yu Li, Bachelor, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine; Qin yang Liu, Bachelor, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine
Locations (1):
- Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing, China

IPD SHARING:
Plan to Share IPD: No